CLINICAL TRIAL: NCT03072173
Title: The Role of the Nose in Snoring and Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: LovisenbergH
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-02

CONDITIONS: Nasal Obstruction; Apnea, Obstructive Sleep
MeSH Terms: conditions — Nasal Obstruction; Sleep Apnea, Obstructive | interventions — xylometazoline; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSG with Xylometazoline then placebo (Experimental): Patients are administered nasal CPAP with humidifier prior to PSG
  Patients in this arm receive Xylometazoline on night 2 of PSG and placebo on night 3 of PSG.
  Interventions: Drug: Xylometazoline; Drug: placebo (saline)
- PSG with placebo then Xylometazoline (Experimental): Patients are administered nasal CPAP with humidifier prior to PSG
  Patients in this arm receive placebo on night 2 of PSG and Xylometazoline on night 3 of PSG.
  Interventions: Drug: Xylometazoline; Drug: placebo (saline)

INTERVENTIONS:
Drug: Xylometazoline — Patient will be given a nasal decongestant (Xylometazoline) prior to their 2nd or 3rd night of PSG.
Drug: placebo (saline) — Patient will be given a placebo nasal spray (saline) prior to their 2nd or 3rd night of PSG.

SUMMARY:
We intend to study, in depth, the quantitative and qualitative properties of nasal respiration in sleep-disordered breathing and sleep apnea and its relation to (CPAP) treatment with the final goal of improving patient outcome.

To do this we will temporarily alter patients' nasal airflow during monitored sleep to lower CPAP air pressure, making CPAP treatment more acceptable to the patient. Additionally we plan to implement highly advanced computerized modelling in collaboration with the OSASMOD research consortium at St. Olavs Hospital/NTNU and SINTEF to predict the results of our alterations and ultimately, to use these predictions to improve both the planning and the outcomes of nasal surgery.

DETAILED DESCRIPTION:
Based on results from previous studies we hypothesize that the nose plays a more significant role in normal sleep respiration and in particular a larger role in sleep disordered breathing than previously recorded.

The overall aim of this project is to gain insight into nasal respiration during wake and sleep, its anatomy, physiology and pathophysiology.

Additionally, we will look at olfactory dysfunction, or reduced sense of smell, a known problem in OSAS patients (n=30), and try to determine if this dysfunction has to do with disturbed sleep architecture or as a result of frequent deoxygenations during the night.

To do this we propose to implement current diagnostic tools available in the diagnostics of sleep disordered breathing such as polysomnography (PSG), in combination with rhinological investigations with 4-phase rhinomanometry and techniques such as two-way fluid structure interaction (FSI) computational fluid dynamic (CFD) analysis of patients. For olfactory testing we will use standardized smell tests. These examinations in combination will give us a more detailed view of the factors that influence nasal respiration.

Additionally, we will use an interventional approach in the proposed study. Patient nasal resistance will be modified under monitored sleep by implementing conventional decongestant nasal spray in an double blinded RCT in order to study the effect of varying nasal resistance on nocturnal respiration and sleep architecture.

Findings, where applicable, will be compared with two-way fluid structure interaction computational fluid dynamic models of patients in all studies to find correlative values and thus assess the predicative value of such computer models.

In the short term these findings could improve patient adherence to CPAP by lowering CPAP pressure. Long term aims are to improve the accuracy of nasal surgery.

Potential end points in our research are as follows:

A better understanding of nasal respiration as a whole Better treatment adherence and satisfaction in sleep apnea patients Improved treatment strategies for sleep apnea patients Improved diagnostics of nasal airflow pathology More focused targeting of medical and surgical intervention in impaired nasal airflow

ELIGIBILITY:
Inclusion Criteria:

* Patients with manifest OSAS and in need of CPAP-treatment

Exclusion Criteria:

* Not speaking Norwegian Language, Congestive heart failure (ejection fraction <40%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Level in therapeutic CPAP pressure | 6 months
  Therapeutic CPAP pressure levels are measured automatically in CPAP device

CONTACTS AND LOCATIONS:
Overall Officials: Søren Berg, MD PhD, Study Chair — University of Lund
Locations (1):
- Lovisenberg Diaconal Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoel HC, Kvinnesland K, Berg S. Outcome of nasal measurements in patients with OSA - Mounting evidence of a nasal endotype. Sleep Med. 2023 Mar;103:131-137. doi: 10.1016/j.sleep.2023.01.028. Epub 2023 Feb 3. PMID 36791622
- [Derived] Hoel HC, Kvinnesland K, Berg S. Impact of nasal resistance on the distribution of apneas and hypopneas in obstructive sleep apnea. Sleep Med. 2020 Jul;71:83-88. doi: 10.1016/j.sleep.2020.03.024. Epub 2020 Apr 17. PMID 32502854